CLINICAL TRIAL: NCT00409058
Title: An Online Intervention for Families Following Adolescent TBI - Teen Online Problem Solving (TOPS)
Brief Title: Teen Online Problem Solving (TOPS) - An Online Intervention Following TBI
Acronym: TOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 05-10-36; H133G050239 (Other Grant/Funding Number: NIDRR)
Record Dates: First submitted 2006-12-07; First posted 2006-12-08 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-09

CONDITIONS: TBI (Traumatic Brain Injury); Brain Edema; Craniocerebral Trauma; Hematoma; Brain Concussion
Keywords: TBI (Traumatic Brain Injury); Intracranial Edema; Brain Edema; Craniocerebral Trauma; Head Injury; Brain Hemorrhage, Traumatic; Subdural Hematoma; Brain Concussion; Head Injuries, Closed
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Edema; Craniocerebral Trauma; Hematoma; Brain Concussion; Brain Hemorrhage, Traumatic; Hematoma, Subdural; Head Injuries, Closed | interventions — TOPS

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teen Online Problem Solving (Experimental): The TOPS program has 10 sessions that provide training in stress management, problem solving, communication, and social skills to all enrolled families, while the remaining 6 sessions address content related to the stressors and burdens of individual families. Each self-guided online session includes real adolescents talking about how TBI affected them, content regarding the skill, video clips showing adolescents and/or families modeling the skill, and exercises giving the family an opportunity to practice the skill. After the completion of the self-guided web pages, the family will meet with the therapist via videoconference; the therapist will review the exercises and help the family implement the problem-solving process with a problem or goal identified by the family.
  Interventions: Behavioral: Teen Online Problem Solving
- Internet Resources Comparison (Experimental): Families in the IRC group will also receive a computer, printer, and high-speed internet access if they do not currently have these. Additionally, IRC families receive access to a home page of brain injury resources and links (identical to those given on the TOPS and TOPS-TO homepage) but will not be able to access specific session content. This will enable us to equate the groups with respect to access to the information and resources available on the Web.
  Interventions: Behavioral: Teen Online Problem Solving

INTERVENTIONS:
Behavioral: Teen Online Problem Solving — We will test the following hypotheses: 1) Children with TBI receiving TOPS will have fewer behavior problems, greater social competence, and better functioning than those receiving IRC at both post-treatment and at a 6-month follow-up assessment. 2) Caregivers of children receiving TOPS will report less depression and psychological distress, less parent-child conflict, and better family functioning than those receiving IRC at both post-treatment and at a 6-month follow-up assessment. 3) Social resources will moderate treatment efficacy, such that children with limited social and economic resources will show greater improvements in the more comprehensive TOPS intervention. We hypothesize better teen problem solving and communication skills, fewer teen emotional/behavioral problems, less parental burden and distress, and less parent-teen conflict at follow-up among the TOPS group compared to the IRC group.
  Other Names: TOPS; IRC

SUMMARY:
The purpose of this study is to learn if using the World Wide Web to train teens and their families in problem-solving, communication skills, and stress management strategies can help them to cope better following traumatic brain injury (TBI). To answer this question, we will look at changes from before the intervention to after the intervention on questionnaire measures of problem-solving skills, communication, social competence, adjustment, and family stress and burden. We hypothesize that families receiving the TOPS intervention will have better parent-child communication and problem-solving skills at follow-up than those receiving the IRC intervention. Additionally, families receiving the TOPS intervention will have lower levels of parental distress, fewer child behavior problems and better child functioning than those receiving the IRC intervention. Lastly, treatment effects will be moderated by SES and life stresses, such that families with greater social disadvantage will benefit more from the TOPS intervention.

DETAILED DESCRIPTION:
Traumatic Brain Injury (TBI) creates significant stress for families resulting in increased burden, anxiety and depression among family members. Both pre- and post-injury family functioning have been linked to child outcomes, suggesting that improvements in family adaptation may result in fewer social and behavioral sequelae in the injured child. Despite this evidence, the development and evaluation of family interventions following TBI are extremely rare.

Children with TBI are often treated at urban trauma centers then discharged to distant home communities where psychosocial follow-up is limited and/or difficult to access. Increasingly, the World Wide Web is being used to meet the mental and other health needs of individuals who have difficulty accessing care through traditional routes. Given the lack of specialized care and follow-up for TBI in many communities, the Web may provide an invaluable tool for linking families with state-of-the-art psychosocial care by reducing potential physical and psychological barriers (e.g., distance, stigma).

Building on previous intervention research of the PI, this study targets the adolescent population between the ages of 12-18. By identifying the unique concerns and issues of this population following brain injury, Teen Online Problem Solving seeks to improve family and teen adaptation, thereby reducing social and behavioral sequelae.

Comparison(s): Teen Online Problem Solving (TOPS) intervention with online curriculum and sequential videoconference therapy sessions in addition to usual care, compared to Internet Resource Comparison with online access to resources in addition to usual care.

ELIGIBILITY:
Inclusion Criteria:

* between 11 and 18 years of age
* moderate to severe traumatic brain injury
* overnight hospital stay
* injury occurred within the last 12 months

Exclusion Criteria:

* younger than 11 and older than 18 years of age
* injury occurred more than 12 months ago
* teen does not live with parents or guardian
* English not spoken in the home
* injury is a result of child abuse as documented by medical record
* child or parent has history of hospitalization for a psychiatric problem
* documentation that the injury is a result of child abuse
* child suffered a non-blunt injury (e.g. projectile wounds, stroke, drowning, or other form of asphyxiation)
* child ever diagnosed with moderate or severe mental retardation, Autism, or a significant developmental disability (child must be able to talk)
* plans for the child to leave home during the coming 12 months.

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2005-10; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Parent Report Measures | 4 years

SECONDARY OUTCOMES:
Teen Self-Report Measures | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Shari L Wade, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (2):
- United States (2):
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio

REFERENCES:
- [Derived] Wade SL, Fisher AP, Kaizar EE, Yeates KO, Taylor HG, Zhang N. Recovery Trajectories of Child and Family Outcomes Following Online Family Problem-Solving Therapy for Children and Adolescents after Traumatic Brain Injury. J Int Neuropsychol Soc. 2019 Oct;25(9):941-949. doi: 10.1017/S1355617719000778. Epub 2019 Aug 13. PMID 31405391
- [Derived] Wade SL, Kaizar EE, Narad M, Zang H, Kurowski BG, Yeates KO, Taylor HG, Zhang N. Online Family Problem-solving Treatment for Pediatric Traumatic Brain Injury. Pediatrics. 2018 Dec;142(6):e20180422. doi: 10.1542/peds.2018-0422. Epub 2018 Nov 9. PMID 30413559
- [Derived] Wade SL, Walz NC, Carey J, McMullen KM, Cass J, Mark E, Yeates KO. A randomized trial of teen online problem solving: efficacy in improving caregiver outcomes after brain injury. Health Psychol. 2012 Nov;31(6):767-76. doi: 10.1037/a0028440. Epub 2012 Jul 2. PMID 22746261